CLINICAL TRIAL: NCT01082874
Title: A Large, International, Placebo-controlled, Factorial Trial to Assess the Impact of Clonidine and Acetyl-salicylic Acid (ASA) in Patients Undergoing Noncardiac Surgery Who Are at Risk of a Perioperative Cardiovascular Event
Brief Title: PeriOperative ISchemic Evaluation-2 Trial
Acronym: POISE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POISE-2 01MAR2010; 2009-018173-31 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Cardiovascular Disease
Keywords: Randomized Controlled Trial; Blinded; Clonidine; acetyl-salicylic acid (ASA); Perioperative vascular complications; Noncardiac surgery
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Clonidine; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active Clonidine and Active ASA (Experimental)
  Interventions: Drug: Active Clonidine; Drug: Active ASA
- Active Clonidine and Placebo ASA (Experimental)
  Interventions: Drug: Active Clonidine; Drug: Placebo ASA
- Placebo Clonidine and Active ASA (Experimental)
  Interventions: Drug: Placebo Clonidine; Drug: Active ASA
- Placebo Clonidine and Placebo ASA (Placebo Comparator)
  Interventions: Drug: Placebo Clonidine; Drug: Placebo ASA

INTERVENTIONS:
Drug: Active Clonidine — Pre-op (goal 2-4 hours): 2 x 0.1mg oral tablets and transdermal patch (0.2 mg/day). Patch to be removed 72 hours post-op.
  Other Names: CATAPRES, CATAPRES-TTS
  Arms: Active Clonidine and Active ASA; Active Clonidine and Placebo ASA
Drug: Placebo Clonidine — Pre-op (goal 2-4 hours): 2 oral placebo tablets and transdermal placebo patch. Patch to be removed 72 hours post-op.
  Arms: Placebo Clonidine and Active ASA; Placebo Clonidine and Placebo ASA
Drug: Active ASA — Pre-op (goal 2-4 hours): 2 x 100mg oral tablets. Post-op: patients ingest one tablet a day (100 mg ASA) for 7 days if patient was were taking ASA chronically prior to surgery or for 30 days if they were not chronically taking ASA prior to surgery
  Other Names: ASPIRIN
  Arms: Active Clonidine and Active ASA; Placebo Clonidine and Active ASA
Drug: Placebo ASA — Pre-op (goal 2-4 hours): 2 oral placebo tablets. Post-op: patients ingest one placebo tablet a day for 7 days if patient was were taking ASA chronically prior to surgery or for 30 days if they were not chronically taking ASA prior to surgery
  Arms: Active Clonidine and Placebo ASA; Placebo Clonidine and Placebo ASA

SUMMARY:
Major surgeries not involving the heart are common, and major heart problems during or after such surgeries represent a large population health problem. Few treatments to prevent heart problems around the time of surgery have been tested. There is encouraging data suggesting that small doses of Acetyl-Salicylic Acid (ASA) and Clonidine, which are two medications, given individually for a short period before and after major surgeries may prevent major heart problems. The POISE-2 Trial is a large international study to test if ASA and Clonidine can prevent heart attacks and deaths from heart problems around the time of surgery.

DETAILED DESCRIPTION:
POISE-2 is a multicentre, international, blinded, 2x2 factorial randomized controlled trial of acetyl-salicylic acid (ASA) and clonidine. The primary objective is to determine the impact of clonidine versus placebo and ASA versus placebo on the 30-day risk of all-cause mortality or nonfatal myocardial infarction in patients with, or at risk of, atherosclerotic disease who are undergoing noncardiac surgery. Patients in the POISE-2 trial will be randomly assigned to one of four groups: ASA and Clonidine together, ASA and Clonidine placebo, ASA placebo and Clonidine, or a ASA placebo and Clonidine placebo. Research personnel will follow patients at 30 days post-randomization and 1 year post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Are undergoing noncardiac surgery;
2. Are ≥ 45 years of age;
3. Are expected to require at least an overnight hospital admission after surgery; AND
4. Fulfill one or more of the following 5 criteria:

   * History of coronary artery disease
   * History of peripheral vascular disease
   * History of stroke
   * Undergoing major vascular surgery
   * Any 3 of the following 9 criteria:

     * undergoing major surgery (i.e. intraperitoneal, intrathoracic, retroperitoneal or major orthopedic surgery
     * history of congestive heart failure
     * transient ischemic attack
     * diabetes and currently taking an oral hypoglycemic agent or insulin
     * age ≥ 70 years
     * hypertension
     * serum creatinine > 175 µmol/L (> 2.0 mg/dL)
     * history of smoking within 2 years of surgery
     * undergoing urgent/emergent surgery

Exclusion Criteria:

1. Consumption of ASA within 72 hours prior to surgery
2. Hypersensitivity or known allergy to ASA or clonidine
3. Systolic blood pressure < 105 mm Hg
4. Heart rate < 55 beats per minute in a patient who does not have a permanent pacemaker
5. Second or third degree heart block without a permanent pacemaker
6. Active peptic ulcer disease or gastrointestinal bleeding within previous 6 weeks
7. Intracranial hemorrhage documented by neuro-imaging, in the 6 months prior to randomization. This does not include petechial hemorrhagic transformation of a primary ischemic stroke
8. Subarachnoid hemorrhage or epidural hematoma unless the event occurred more than 6 months prior to randomization and the offending aneurysm or arterial lesion has been repaired
9. Drug-eluting coronary stent in the year prior to randomization
10. Bare-metal coronary stent in the 6 weeks prior to randomization
11. Thienopyridine (e.g., clopidogrel, ticlopidine, prasugrel) or ticagrelor within 72 hours prior to surgery; or intent to restart a thienopyridine or ticagrelor during the first 7 days post-op; or currently taking an alpha-2 agonist, alpha methyldopa, monoamine oxidase inhibitors or reserpine;
12. Planned use - during the first 3 days after surgery - therapeutic dose anticoagulation or a therapeutic subcutaneous or intravenous antithrombotic agent
13. Undergoing intracranial surgery, carotid endarterectomy, or retinal surgery
14. Not consenting to participate in POISE-2 prior to surgery
15. Previously enrolled in POISE-2 Trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10010 (Actual)
Dates: Start 2010-07; Primary Completion 2014-03 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P.J. Devereaux, MD, PhD, Principal Investigator — Population Health Research Institute; Salim Yusuf, DPhil, Study Chair — Population Health Research Institute
Locations (23):
- National Coordination Office, Cleveland, Ohio, United States
- National Coordination Office, Rosario, Argentina
- National Coordination Office Australia and New Zealand, Parkville, Victoria, Australia
- National Coordination Office, Vienna, Austria
- National Coordination Office, Brussels, Belgium
- National Coordination Office, São Paulo, Brazil
- National Coordination Office, Hamilton, Ontario, Canada
- National Coordination Office, Santiago, Chile
- National Coordination Office, Bucamaranga, Colombia
- National Coordination Office, Herlev, Denmark
- National Coordination Office, Boulogne-Billancourt, France
- National Coordination Office, Bonn, Germany
- National Coordination Office, Hong Kong, Hong Kong
- National Coordination Office, Bangalore, India
- National Coordination Office, Milan, Italy
- National Coordination Office, Kuala Lumpur, Malaysia
- National Coordination Office, Auckland, New Zealand
- National Coordination Office, Islamabad, Pakistan
- National Coordination Office, Lima, Peru
- National Coordination Office, Durban, South Africa
- National Coordination Office, Barcelona, Spain
- National Coordination Office, Basel, Switzerland
- National Coordination Office, Hull, United Kingdom

REFERENCES:
- [Result] Devereaux PJ, Mrkobrada M, Sessler DI, Leslie K, Alonso-Coello P, Kurz A, Villar JC, Sigamani A, Biccard BM, Meyhoff CS, Parlow JL, Guyatt G, Robinson A, Garg AX, Rodseth RN, Botto F, Lurati Buse G, Xavier D, Chan MT, Tiboni M, Cook D, Kumar PA, Forget P, Malaga G, Fleischmann E, Amir M, Eikelboom J, Mizera R, Torres D, Wang CY, VanHelder T, Paniagua P, Berwanger O, Srinathan S, Graham M, Pasin L, Le Manach Y, Gao P, Pogue J, Whitlock R, Lamy A, Kearon C, Baigent C, Chow C, Pettit S, Chrolavicius S, Yusuf S; POISE-2 Investigators. Aspirin in patients undergoing noncardiac surgery. N Engl J Med. 2014 Apr 17;370(16):1494-503. doi: 10.1056/NEJMoa1401105. Epub 2014 Mar 31. PMID 24679062
- [Result] Devereaux PJ, Sessler DI, Leslie K, Kurz A, Mrkobrada M, Alonso-Coello P, Villar JC, Sigamani A, Biccard BM, Meyhoff CS, Parlow JL, Guyatt G, Robinson A, Garg AX, Rodseth RN, Botto F, Lurati Buse G, Xavier D, Chan MT, Tiboni M, Cook D, Kumar PA, Forget P, Malaga G, Fleischmann E, Amir M, Eikelboom J, Mizera R, Torres D, Wang CY, Vanhelder T, Paniagua P, Berwanger O, Srinathan S, Graham M, Pasin L, Le Manach Y, Gao P, Pogue J, Whitlock R, Lamy A, Kearon C, Chow C, Pettit S, Chrolavicius S, Yusuf S; POISE-2 Investigators. Clonidine in patients undergoing noncardiac surgery. N Engl J Med. 2014 Apr 17;370(16):1504-13. doi: 10.1056/NEJMoa1401106. Epub 2014 Mar 31. PMID 24679061
- [Result] Garg AX, Kurz A, Sessler DI, Cuerden M, Robinson A, Mrkobrada M, Parikh C, Mizera R, Jones PM, Tiboni M, Rodriguez RG, Popova E, Rojas Gomez MF, Meyhoff CS, Vanhelder T, Chan MT, Torres D, Parlow J, de Nadal Clanchet M, Amir M, Bidgoli SJ, Pasin L, Martinsen K, Malaga G, Myles P, Acedillo R, Roshanov P, Walsh M, Dresser G, Kumar P, Fleischmann E, Villar JC, Painter T, Biccard B, Bergese S, Srinathan S, Cata JP, Chan V, Mehra B, Leslie K, Whitlock R, Devereaux PJ; POISE-2 Investigators. Aspirin and clonidine in non-cardiac surgery: acute kidney injury substudy protocol of the Perioperative Ischaemic Evaluation (POISE) 2 randomised controlled trial. BMJ Open. 2014 Feb 25;4(2):e004886. doi: 10.1136/bmjopen-2014-004886. PMID 24568963
- [Derived] Roshanov PS, Walsh MW, Garg AX, Cuerden M, Lam NN, Hildebrand AM, Lee VW, Mrkobrada M, Leslie K, Chan MTV, Borges FK, Wang CY, Xavier D, Sessler DI, Szczeklik W, Meyhoff CS, Srinathan SK, Sigamani A, Villar JC, Chow CK, Polanczyk CA, Patel A, Harrison TG, Fielding-Singh V, Cata JP, Parlow J, de Nadal M, Devereaux PJ. Preoperative estimated glomerular filtration rate to predict cardiac events in major noncardiac surgery: a secondary analysis of two large international studies. Br J Anaesth. 2025 Feb;134(2):297-307. doi: 10.1016/j.bja.2024.10.039. Epub 2025 Jan 2. PMID 39753401
- [Derived] Turan A, Rivas E, Devereaux PJ, Pu X, Rodriguez-Patarroyo FA, Yalcin EK, Nault R, Maheshwari K, Ruetzler K, Sessler DI. Relative contributions of anaemia and hypotension to myocardial infarction and renal injury: Post hoc analysis of the POISE-2 trial. Eur J Anaesthesiol. 2023 May 1;40(5):365-371. doi: 10.1097/EJA.0000000000001816. Epub 2023 Mar 9. PMID 36891761
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Biccard BM, Sigamani A, Chan MTV, Sessler DI, Kurz A, Tittley JG, Rapanos T, Harlock J, Szalay D, Tiboni ME, Popova E, Vasquez SM, Kabon B, Amir M, Mrkobrada M, Mehra BR, El Beheiry H, Mata E, Tena B, Sabate S, Zainal Abidin MK, Shah VR, Balasubramanian K, Devereaux PJ. Effect of aspirin in vascular surgery in patients from a randomized clinical trial (POISE-2). Br J Surg. 2018 Nov;105(12):1591-1597. doi: 10.1002/bjs.10925. Epub 2018 Jul 18. PMID 30019751
- [Derived] Graham MM, Sessler DI, Parlow JL, Biccard BM, Guyatt G, Leslie K, Chan MTV, Meyhoff CS, Xavier D, Sigamani A, Kumar PA, Mrkobrada M, Cook DJ, Tandon V, Alvarez-Garcia J, Villar JC, Painter TW, Landoni G, Fleischmann E, Lamy A, Whitlock R, Le Manach Y, Aphang-Lam M, Cata JP, Gao P, Terblanche NCS, Ramana PV, Jamieson KA, Bessissow A, Mendoza GR, Ramirez S, Diemunsch PA, Yusuf S, Devereaux PJ. Aspirin in Patients With Previous Percutaneous Coronary Intervention Undergoing Noncardiac Surgery. Ann Intern Med. 2018 Feb 20;168(4):237-244. doi: 10.7326/M17-2341. Epub 2017 Nov 14. PMID 29132159
- [Derived] Garg AX, Kurz A, Sessler DI, Cuerden M, Robinson A, Mrkobrada M, Parikh CR, Mizera R, Jones PM, Tiboni M, Font A, Cegarra V, Gomez MF, Meyhoff CS, VanHelder T, Chan MT, Torres D, Parlow J, Clanchet Mde N, Amir M, Bidgoli SJ, Pasin L, Martinsen K, Malaga G, Myles P, Acedillo R, Roshanov PS, Walsh M, Dresser G, Kumar P, Fleischmann E, Villar JC, Painter T, Biccard B, Bergese S, Srinathan S, Cata JP, Chan V, Mehra B, Wijeysundera DN, Leslie K, Forget P, Whitlock R, Yusuf S, Devereaux PJ; POISE-2 Investigators. Perioperative aspirin and clonidine and risk of acute kidney injury: a randomized clinical trial. JAMA. 2014 Dec 3;312(21):2254-64. doi: 10.1001/jama.2014.15284. PMID 25399007
- [Derived] Devereaux PJ; POISE-2 Investigators. Rationale and design of the PeriOperative ISchemic Evaluation-2 (POISE-2) trial: an international 2 x 2 factorial randomized controlled trial of acetyl-salicylic acid vs. placebo and clonidine vs. placebo in patients undergoing noncardiac surgery. Am Heart J. 2014 Jun;167(6):804-9.e4. doi: 10.1016/j.ahj.2014.01.007. Epub 2014 Feb 22. PMID 24890528
- [Derived] Chludzinski A, Irani C, Mascha EJ, Kurz A, Devereaux PJ, Sessler DI. Protocol understanding and anxiety in perioperative clinical trial patients approached for consent on the day of surgery. Mayo Clin Proc. 2013 May;88(5):446-54. doi: 10.1016/j.mayocp.2012.12.014. PMID 23639498

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Clonidine and Active ASA | Active Clonidine and Placebo ASA | Placebo Clonidine and Active ASA | Placebo Clonidine and Placebo ASA
Started | 2499 | 2510 | 2499 | 2502
Completed | 2488 | 2498 | 2488 | 2489
Not Completed | 11 | 12 | 11 | 13
Not completed — Lost to Follow-up | 10 | 10 | 6 | 10
Not completed — Withdrawal by Subject | 1 | 2 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Clonidine and Active ASA | Active Clonidine and Placebo ASA | Placebo Clonidine and Active ASA | Placebo Clonidine and Placebo ASA | Total
Number analyzed (Participants) | 2499 | 2510 | 2499 | 2502 | 10010
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 873 | 836 | 836 | 866 | 3411
  >=65 years | 1626 | 1674 | 1663 | 1636 | 6599
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.4) | 68.6 (10.3) | 68.7 (10.2) | 68.5 (10.3) | 68.6 (10.3)
Gender [Number; unit: participants]
  Female | 1212 | 1164 | 1188 | 1160 | 4724
  Male | 1287 | 1346 | 1310 | 1340 | 5283
Region of Enrollment [Number; unit: participants]
  Colombia | 162 | 161 | 164 | 162 | 649
  Argentina | 3 | 2 | 3 | 3 | 11
  Hong Kong | 69 | 70 | 69 | 68 | 276
  United States | 443 | 440 | 437 | 440 | 1760
  United Kingdom | 22 | 22 | 22 | 20 | 86
  Malaysia | 30 | 28 | 30 | 32 | 120
  Switzerland | 24 | 24 | 25 | 23 | 96
  India | 149 | 149 | 151 | 146 | 595
  Spain | 133 | 139 | 131 | 135 | 538
  New Zealand | 14 | 11 | 11 | 10 | 46
  Canada | 875 | 878 | 872 | 873 | 3498
  Austria | 44 | 44 | 42 | 46 | 176
  Pakistan | 43 | 44 | 44 | 44 | 175
  Belgium | 44 | 47 | 46 | 47 | 184
  Brazil | 13 | 12 | 16 | 16 | 57
  Denmark | 80 | 80 | 80 | 81 | 321
  Italy | 39 | 39 | 38 | 38 | 154
  South Africa | 87 | 87 | 89 | 90 | 353
  Australia | 119 | 120 | 113 | 118 | 470
  Chile | 38 | 38 | 38 | 39 | 153
  France | 21 | 24 | 24 | 20 | 89
  Peru | 41 | 44 | 43 | 44 | 172
  Germany | 6 | 7 | 11 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Composite of All-cause Mortality and Nonfatal MI
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Active Clonidine and Active ASA | Active Clonidine and Placebo ASA | Placebo Clonidine and Active ASA | Placebo Clonidine and Placebo ASA
Number analyzed (Participants) | 2499 | 2510 | 2499 | 2502
participants | 173 | 194 | 178 | 161

2. Primary Outcome: All-cause Mortality and Nonfatal MI
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Composite of All-cause Mortality, Nonfatal MI, and Nonfatal Stroke
Time Frame: 30 days
Reporting Status: Not Posted

4. Secondary Outcome: Individual Secondary Outcomes
Description: All-cause mortality, vascular mortality, MI, nonfatal cardiac arrest, cardiac revascularization procedure, pulmonary emboli, deep venous thrombosis, clinically important atrial fibrillation, amputation, peripheral arterial thrombosis, infection/sepsis, rehospitalization for vascular reasons, length of hospital stay, length of intensive care unit / cardiac care unit (ICU/CCU) stay, and new acute renal failure requiring dialysis.
Time Frame: 30 days
Reporting Status: Not Posted

5. Secondary Outcome: Composite Outcome by ASA Stratum
Description: Composite outcome of all-cause mortality, nonfatal MI, cardiac revascularization procedure, nonfatal pulmonary emboli, and nonfatal deep venous thrombosis.
Time Frame: 30 days
Reporting Status: Not Posted

6. Secondary Outcome: Safety Outcomes in ASA Trial
Description: Stroke, congestive heart failure, life-threatening bleeding, and major bleeding.
Time Frame: 30 days
Reporting Status: Not Posted

7. Secondary Outcome: Safety Outcomes in Clonidine Trial
Description: Stroke, clinically important hypotension, clinically important bradycardia, and congestive heart failure.
Time Frame: 30 days
Reporting Status: Not Posted

8. Secondary Outcome: Composite Outcome at 1 Year
Description: All-cause mortality, nonfatal MI, and nonfatal stroke.
Time Frame: 1 year
Reporting Status: Not Posted

9. Secondary Outcome: Individual Secondary Outcomes at 1 Year
Description: All cause mortality, vascular mortality, MI, nonfatal cardiac arrest, cardiac revascularization procedure, stroke, pulmonary emboli, deep venous thrombosis, amputation, peripheral arterial thrombosis, new diagnosis of cancer, diagnosis of recurrent cancer and rehospitalization for vascular reason.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Active Clonidine and Active ASA | Active Clonidine and Placebo ASA | Placebo Clonidine and Active ASA | Placebo Clonidine and Placebo ASA
Serious Adverse Events (participants affected / at risk) | 46/2499 | 52/2510 | 45/2499 | 39/2502
Other Adverse Events (participants affected / at risk) | 0/2499 | 0/2510 | 0/2499 | 0/2502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Clonidine and Active ASA (N=2499) | Active Clonidine and Placebo ASA (N=2510) | Placebo Clonidine and Active ASA (N=2499) | Placebo Clonidine and Placebo ASA (N=2502)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dissemianted intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachy Arrythymia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Open Angle Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterovesicle Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI Hemmorhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernial Eventration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Intestinal Dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Fistuala (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Ischemia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumoretroperitonium (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectum hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Samll Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Device Dislocation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired Healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ Failure (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischemic Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Wound Dehisence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endotrachial Intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fascial Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Stoma Necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerous Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision Site Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Lymphatic Duct Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound Evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wound Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Systolic Increase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decrease (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Internatinal Normalized Ratio Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver Functin Test Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracic Cavity Drainage test Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
b-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine Carcinoma Metatastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peroneal Nerve Palsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pre-syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
TIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0
Vasculitis Cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vocal Cord Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusinal State (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dilirium (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Emotional Distress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Pre-renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic-UretericObstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Cyst Rupture (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Renal Ischemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actue Respiratory Distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Broncho Spasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lymphorrhoea (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No